CLINICAL TRIAL: NCT05358431
Title: Stratification of Presymptomatic Amyotrophic Lateral Sclerosis: the Development of Novel Imaging Biomarkers
Acronym: STRATALS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP211449; 2022-A00083-40 (Other: IDRCB)
Record Dates: First submitted 2022-02-17; First posted 2022-05-03 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: MRI; ALS; FTD; MUNE; C9orfF72; presymptomatic
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Neuroimaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- participants (Experimental): Patients fulfilling the El Escorial criteria for probable or definite ALS with a C9orf72 mutation or asymptomatics being a first-degree to a person carrying a C9orf72 mutation or Healthy controls
  Interventions: Other: Neuroimaging and electrophysiology

INTERVENTIONS:
Other: Neuroimaging and electrophysiology — Brain and spinal cord MRI, transcranial magnetic stimulation; Motor Unit Number Estimation, EEG

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a relentlessly progressive neurodegenerative disorder with no effective disease-modifying therapies at present. The disease is sporadic in 90 % of the ALS patients. Up to 40 % familial ALS cases and up to 25% of familial frontotemporal dementia (FTD) are caused by autosomal dominant GGGGCC hexanucleotide repeat expansions in the C9orf72 gene. The presymptomatic phase of the disease represents a unique opportunity to evaluate mechanisms of disease propagation, characterise patterns of anatomical spread, validate staging systems and appraise the comparative sensitivity profile of emerging imaging modalities. Very few spinal cord imaging studies currently exist in ALS despite their potential to characterise both the lower and upper motor neuron components of the disease. This prospective longitudinal study of asymptomatic and symptomatic c9orf72 hexanucleotide carriers will use a purpose-designed spinal and brain imaging protocol and comprehensive clinical, genetic, electrophysiological and neuropsychological profiling. Newly developed imaging techniques such as spinal cord NODDI, spinal fMRI, quantitative thoracic cord imaging will be implemented in addition to established spinal cord and brain imaging techniques.

DETAILED DESCRIPTION:
The main objective is to study the disease trajectory from the presymptomatic to the symptomatic phase of ALS. We will study a population of asymptomatic subjects carrying an autosomal dominant GGGGCC hexanucleotide repeat expansions in the C9orf72 gene that is the most frequent mutation in familial cases of ALS. The changes will be compared to a population of healthy controls. We have selected two populations of healthy controls to take into account the possible interaction with the genetic background. The first population of controls will consist in subjects sharing the same genetic background than the presymptomatic subjects, e.g. non mutated subjects related to C9 + symptomatic carriers. The second population will consist in healthy individuals coming from the general population. We will compare the presymptomatic changes to changes occurring at the symptomatic phase by studying a group of patients with symptomatic ALS. We will use a multimodal longitudinal approach combing spinal and brain imaging protocol and comprehensive clinical, genetic, electrophysiological and neuropsychological profiling.

Secondary objectives

1. Comparison of the changes in young presymptomatic subjects (less than 40 years) vs older patients
2. Changes over time in ALS patients : MRI metrics, electrophysiological parameters and neuropsychological impairment
3. The development of prognostic indicators based on spinal cord/ brain imaging and electrophysiology to foretell phenotypic manifestation (such as DFT or ALS) and age of onset.
4. The integrative evaluation of brain-cord interactions, comparing the relative detection sensitivity of spinal and cerebral imaging measures.
5. Assessing the imaging evidence for the prevailing 'corticofugal spread' or 'dying-forward' theory based on longitudinal spinal cord and cerebral data.
6. Characterizing associations between imaging and electrophysiology metrics of upper motor neuron (UMN) and LMN (lower motor neuron) integrity; correlation of segmental grey matte metrics to MUNIX; TMS to corticospinal tract measures
7. Assessing whether longitudinal cerebral and spinal cord imaging data are consistent with sequential TDP-43 pathological staging systems.
8. The cross-validation of newly developed cord techniques; NODDI, fMRI, thoracic cord imaging with established structural and diffusion imaging metrics and electrophysiology measures.
9. Correlations between imaging, electrophysiology and neuropsychological metrics

ELIGIBILITY:
Inclusion criteria shared by all the different cohorts and controls :

* Age more than 18 years.
* Signature of a consent form for clinical, paraclinical and genetic assessment
* Fluent in French
* Affiliated to the French Security Healthcare System ("Sécurité Sociale")
* Absence of neurological comorbidity (stroke, tumor etc)

The inclusion criteria for asymptomatic relatives :

* Being a first-degree to a person carrying a C9orf72 mutation.
* Absence of proven clinical signs of FTD, ALS, language, praxic, memory disorders, Parkinsonian syndrome.

Inclusion criteria for symptomatic ALS patients :

* Patients fulfilling the El Escorial criteria for probable or definite ALS
* Presence of a C9orf72 mutation

Exclusion criteria for participants from all cohorts :

* Contraindication to MRI and TMS
* Impossibility to stay in decubitus during 1 hour,
* For women, childbearing or breastfeeding
* For women of childbearing potential: positive HCG test or positive urine pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-07-21 (Actual); Primary Completion 2026-02-21 (Estimated); Study Completion 2026-02-21 (Estimated)

PRIMARY OUTCOMES:
Functional and structural quantitative imaging | 6 months
  Changes in resting state spinal cord MRI (fMRI) signal in presymptomatic and symptomatic ALS patients compared to controls

SECONDARY OUTCOMES:
Electromyography with MUNE | 6 months
  Difference between electrophysiological MUNE between the first and last visit
TMS | 6 months
  Difference between electrophysiological TMS between the first and last visit
EEG | 6 months
  Difference between electrophysiological "Resting state (rs-)EEG" ,alpha (7-13 Hz), beta (13-40 Hz) and gamma bands (40-200 Hz) between the first and last visit

CONTACTS AND LOCATIONS:
Locations (1):
- ICM, GH Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saracino D, Cipriano L, Houot M, Querin G, Rinaldi D, Rametti-Lacroux A, Wallon D, Gerardin E, Couratier P, Boncoeur MP, Lebouvier T; PREV-DEMALS and STRATALS study groups; Colliot O, Pradat PF, Migliaccio R, Le Ber I. Quantifying multimodal longitudinal brain changes in presymptomatic C9orf72 disease. Alzheimers Dement. 2025 Dec;21(12):e70902. doi: 10.1002/alz.70902. PMID 41366786